CLINICAL TRIAL: NCT00514865
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of ONO-2333Ms in Patients With Recurrent Major Depressive Disorder
Brief Title: Placebo-Controlled Study of ONO-2333Ms in Patients With Recurrent Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-2333POU007
Record Dates: First submitted 2007-08-07; First posted 2007-08-10 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: ONO-2333Ms; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Experimental 1 (Experimental): 1-2 mg of ONO-2333
  Interventions: Drug: ONO-2333Ms Experimental 1
- Experimental 2 (Experimental): 5-10 mg of ONO-2333
  Interventions: Drug: ONO-2333Ms Experimental 2
- Placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2333Ms Experimental 2 — 5-10 mg QD(once a day) for 8 weeks
  Arms: Experimental 2
Drug: Placebo — 0 mg QD(once a day) for 8 weeks
  Arms: Placebo
Drug: ONO-2333Ms Experimental 1 — 1-2 mg QD(once a day) for 8 weeks
  Arms: Experimental 1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ONO-2333Ms in patients with Recurrent Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with recurrent major depressive disorder

Exclusion Criteria:

* Patients with treatment resistance for depression
* History of alcohol abuse/dependence, substance abuse/dependence within 6 months
* Has clinically significant unstable medical condition
* Has significant risk of suicide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2007-06-13 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to treatment endpoint in the MADRS total score | 8 weeks

SECONDARY OUTCOMES:
Change from baseline to treatment endpoint in the HAM-D17, QIDS-SR16, CGI-S, CGI-I, PGI score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsutoshi Hatakeyama, M.S., Study Director — Ono Pharma USA Inc
Locations (1):
- Ono Pharma Investigtional Site, Atlanta, Georgia, United States